CLINICAL TRIAL: NCT06147388
Title: Regression of Cervical Precancerous Lesions and Associated Risk Factors
Acronym: RECER
Status: Recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, David Cibula, Dr, PhD, General University Hospital, Prague
Other Study IDs: 154/22 S
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cervix Uteri SIL; HPV; CIN2; CIN3
MeSH Terms: interventions — Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIN 2, CIN 3: Bioptically verified CIN 2 or CIN 3 lesion
  Interventions: Diagnostic Test: Colposcopy

INTERVENTIONS:
Diagnostic Test: Colposcopy — No surgery, observation

SUMMARY:
The aim of this study is to assess the extent of histopathological regression of severe cervical precancerous lesions (CIN 2 and CIN 3); evaluate the proportion of patients who experience the normalization of HPV test and cytology finding among those who were treated conservatively and those who underwent conization; and identify predictive parameters associated with regression. Based on this analysis, a model will be proposed to predict the likelihood of lesion regression.

DETAILED DESCRIPTION:
Introduction There are three grades of dysplasia of the cervix based on their severity (CIN 1-3). Most women with CIN 2 or CIN 3 (high-grade - HG lesions) are referred for conization due to the presumed risk of developing invasive cervical cancer. However, this surgical intervention is associated with an increased risk of preterm labor in the future.

From the literature, it is evident that 30% - 60% of CIN 2 and CIN 3 lesions spontaneously regress. Colposcopic examination is a tool that can accurately assess the severity of the lesion and safely evaluate the dynamics of its development. It can be used to exclude the presence of invasive cervical cancer.

The aim of the study is to determine the absolute rate of spontaneous regression of HG lesions, considering stratification factors.

Methods Patients meeting all inclusion criteria and none of the exclusion criteria are included (see below). Colposcopic evaluations occur at four-month intervals during the study. In case of progression, the patient is indicated for conization; in case of persistence, the patient is consulted and can choose further observation or conization; in case of regression, punch biopsy is performed to acquire a histopathologic sample for primary endpoint evaluation. The biopsy/conization result is subsequently compared with the initial sample to declare regression or persistence of the HG lesion.

The HPV status and cytological findings are evaluated similarly. Stratification criteria such as age, colposcopic characteristics, HPV genotype (Cobas 4800, Roche Molecular Systems, Pleasanton, USA), methylation markers (GynTect®, Oncgnostics GmbH, Löbstedter Str. 41, 07749 Jena, Germany), semiquantitative microscopic assessment of the vaginal swab, and personal history are assessed during monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. squamocolumnar junction fully visualized
2. bioptically verified CIN 2 or CIN 3
3. age ≥ 18 years
4. age ≤ 40 years
5. informed consent

Exclusion Criteria:

1. squamocolumnar junction not fully visualized
2. suspicion on glandular lesion
3. suspicion on invasive cancer
4. personal history of CIN 2, 3 or cerv. cancer
5. gravidity
6. HIV positivity
7. immunosuppression
8. impossible photographic documentation

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Consecutive participant sampling of patients with bioptically-verified CIN 2 or CIN 3 and fully visualised squamocolumnar junction with no suspiction on invasive cancer or glandular lesion.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Regression-rate of severe cervical precancerous lesions (CIN 2 and CIN 3) expressed through a comparison of initial and final histology | 3 years
  Histological results from the initial visit will be compared with the biopsy obtained during the last visit (or the specimen from conization) to determine whether regression or persistence of the high-grade lesion has occurred.

SECONDARY OUTCOMES:
Rate of HPV negativization in patients with spontaneous regression compared to patients with persistence after conization | 3 years
  The proportion of patients with a negative result on the HPV DNA test obtained during the final visit will be assessed.
Rate of cytological normalization in patients with spontaneous regression compared to patients with persistence after conization | 3 years
Regression-rate considering specified stratification factors | 3 years
  Specific factors will be evaluated to determine their influence on the regression or persistence of the cervical high-grade lesion. The following factors will be assessed:
  * CIN Grade (CIN 2 / CIN 3)
  * Immunohistochemically detected biomarkers
  * p16INK4a
  * Ki-67
  * E4
  * Gene methylation (ASTN1, DLX1, ITGA4, RXFP3, SOX17, and ZNF671)
  * Histologically described cervicitis
  * Colposcopic Markers
  * Microbiological Markers
  * Selective HPV genotyping
  * Viral load
  * Anamnestic Data
  * Smoking
  * Age
Development of a model for predicting spontaneous regression | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Prague, Czechia

REFERENCES:
- [Derived] Dostalek L, Brynda D, Marek R, Hederlingova J, Tripac I, Nemejcova K, Slovackova M, Zima T, Cibula D, Slama J. Regression of high-grade squamous intraepithelial cervical lesions and associated risk factors (RECER). Int J Gynecol Cancer. 2025 May;35(5):101768. doi: 10.1016/j.ijgc.2025.101768. Epub 2025 Mar 13. PMID 40215795